CLINICAL TRIAL: NCT04531163
Title: Possible Ameliorating Effect of N- Acetylcysteine on Type-II Diabetes Induced Nephropathy
Brief Title: Possible Ameliorating Effect of N- Acetylcysteine (NAC) on Type-II Diabetes Induced Nephropathy
Acronym: (NAC)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Tasneem Ahmed Hamed, Clinical pharamacist, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AlAzharUn
Record Dates: First submitted 2020-08-21; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Diabetic Kidney Disease; Diabetes Mellitus, Type 2; Diabetic Nephropathies
Keywords: N-Acetyl cysteine; Lipoprotein a; Triglycerides; Total cholesterol; Glycated Haemoglobin; Fasting blood sugar; Serum creatinine; Blood urea nitrogen; Urine analysis; High density lipoprotein; Low density lipoprotein
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2 | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Two arms are being used parallel to each other at the same time. Participants are assigned to two groups in parallel for the duration of the study. One arm is interventional assigned to drug administration and the other is a control arm.
Masking Description: All participants,investigators, care providers, and outcome assessor have knowledge of the interventions assigned to individual participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): First arm is experimental, given (NAC) for 2 months in 1200mg/day dosing.
  Both arms are assigned to pre-treatment analytical tests and post treatment all test analysis are repeated to compare drug effect with placebo group.
  Interventions: Drug: N Acetylcysteine
- Non-interventional (No Intervention): Second arm has no intervention. It is only used to compare results of analytical tests with the first interventional arm.

INTERVENTIONS:
Drug: N Acetylcysteine — (NAC) is a drug used in the experiment and participant are treated with it by 1200mg/day dose for two months.
  Other Names: (NAC); Fluimucil
  Arms: Interventional

SUMMARY:
The study is focused on the possible improving effect of N-acetylcysteine on nephropathy of type-2 diabetic patients.

Study design: Prospective clinical based study. The aim of this work is to study the effect of N-acetylcysteine (NAC) on proteinuria and on the serum level of lipoprotein a (LPa) in diabetes induced nephropathy in type-2 diabetic patients.

DETAILED DESCRIPTION:
This study will be carried on 60 participants with Type 2 Diabetes with age over 20 years.

Participants will be classified into two groups:

1. Group I (Interventional): treated with (NAC) dose of 1200 mg/day for two months in conjunction with conventional treatment.
2. Group II (Non-interventional): control group receive conventional treatment.

All patients will undergo the following:

1. Full medical history will be taken.
2. Laboratory investigations as follows:

Blood samples will be collected for analysis after overnight fasting at the beginning and after 2 months of the study for determination of:

1. Total cholesterol (T-chol).
2. Plasma triglycerides (TG).
3. High density lipoprotein cholesterol (HDL-C).
4. Low density lipoprotein cholesterol (LDL-C).
5. Fasting blood sugar.
6. Blood urea nitrogen (BUN).
7. Serum creatinine (SCr).
8. Urine analysis.
9. Glycated hemoglobin (HbA1c).
10. Lipoprotein (a). In addition, blood pressure will be measured for 24 hr.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of Diabetes Mellitus.
2. Age over 20 years.
3. Patients with proteinuria ≥ 30 mg /dl.

Exclusion Criteria:

1. Patients on lipid lowering medications.
2. Cigarette smokers.
3. Presence of liver and heart diseases.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Lipoprotein (a) | 2 months
  unique lipoprotein that has emerged as an independent risk factor for developing vascular disease.
Triglycerides | 2 months
  Triglycerides are a type of fat (lipid) found in our blood. It is one of the lipid panel used to determine atherosclerotic risk that contributes to vascular diseases.
Systolic blood pressure | 2 months
  The first number of blood pressure reading and it indicates how much pressure our blood is exerting against our artery walls when the heart beats. It is a major risk factor for cardiovascular disease.

CONTACTS AND LOCATIONS:
Overall Officials: Huda M. Salem, PhD, Study Chair — Al-Azhar University
Locations (1):
- Al Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No